CLINICAL TRIAL: NCT01029743
Title: Xarelto® Regulatory Post-Marketing Surveillance
Brief Title: Xarelto Regulatory Post-Marketing Surveillance
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 14793; XA0910KR (Other: company internal)
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Venous Thromboembolism
Keywords: TKR (Total Knee Replacement); THR (Total Hip Replacement); VTE (Venous Thromboembolism); LMWH (Low Molecular Weight Heparin); VKA (Vitamin K antagonist)
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Group 2
  Interventions: Drug: Pharmacologic agents (e.g. LMWH/VKA/Fondaparinux/Aspirin and etc.)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Daily dose, a treatment duration of 5 weeks for patients undergoing major hip surgery and a treatment duration of 2 weeks for patients undergoing major knee surgery are recommended
  Groups: Group 1
Drug: Pharmacologic agents (e.g. LMWH/VKA/Fondaparinux/Aspirin and etc.) — Daily dose, dosage frequency and duration will be decided by physicians
  Groups: Group 2

SUMMARY:
This study is to identify the following problems and questions with respect to the safety and effectiveness of Xarelto in comparison with other pharmacologic agents in the prophylaxis of venous thromboembolism (VTE) in a large sample of patients who undergo elective total hip replacement (THR) or total knee replacement (TKR) in the real-life conditions in its registered indication(s) as required by Korean Food and Drug Administration (KFDA).

1. Known and unknown adverse reactions, especially serious adverse reactions
2. Incidence of adverse reactions under the routine drug use
3. Factors that may affect the safety of the drug
4. Factors that may affect the effectiveness of the drug
5. Other safety information related to overuse, drug interaction and laboratory abnormalities
6. Other adverse reactions

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients >/= 18 years of age who will undergo elective total hip replacement or total knee replacement and receive Xarelto or other pharmacologic standard of care Venous Thromboembolism (VTE) prophylaxis, and who consent to participate in the study

Exclusion Criteria:

* Patients with hypersensitivity to any pharmacologic VTE prophylaxis treatment
* Patients with clinically significant active bleeding (e.g., intracranial bleeding, gastrointestinal bleeding)
* Patients with significant hepatic disease which is associated with coagulopathy leading to a clinically relevant bleeding risk
* Pregnant or lactating women
* Patients with hereditary problems of lactose or galactose intolerance (e.g., the Lapp lactase deficiency or glucose-galactose malabsorption)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be treated with rivaroxaban or other pharmacologic agents (e.g. LMWH/VKA/Fondaparinux) to prevent VTE after elective total hip replacement or total knee replacement
Sampling Method: Non-Probability Sample
Enrollment: 3388 (Actual)
Dates: Start 2009-12; Primary Completion 2015-03 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Adverse event collection | From the start of signed consent to 4 weeks after discharge

SECONDARY OUTCOMES:
Duration of treatment | Whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, South Korea